CLINICAL TRIAL: NCT04506710
Title: Ways to Improve the Efficiency of Communication Between Health Workers and Oncological Patients During Medical Consultative Conversations: an Observational Clinical Study
Brief Title: Improvement of Communicational Skills Between Health Workers and Oncological Patients During Medical Consultative Conversations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Other Study IDs: RSCS-L0838
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with low-risk prostate cancer: Histologically confirmed low-risk prostate cancer (PSA up to 10 ng / ml; Gleason (3 + 3) = 6 (ISUP 1); tumor stage T2a (low- risk according to the D'Amico scale))
  Interventions: Behavioral: Audio recording of the counseling conversation

INTERVENTIONS:
Behavioral: Audio recording of the counseling conversation — The patient will have an audio-recorded counseling conversation. Audio recording will be carried out using a portable recorder ZOOM H2n. The audio recordings of the counseling conversations will be performed by the health workers selected to participate in the study.

SUMMARY:
The aim of the study is to identify the specific patterns of communication between doctors and oncological patients during medical consultations and develop recommendations to improve its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer;
2. PSA up to 10 ng / ml; Gleason (3 + 3) = 6 (ISUP 1); the stage of the tumor T2a (low- risk according to the D'Amico scale);

Exclusion Criteria:

1. Failure of the recording device;
2. Unsatisfactory audio quality.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Males with low-risk prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Identification the communication techniques used by the doctor in the counseling conversation; | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fedorovskaya Viktorya, Study Director — Institute of Linguistics and Intercultural Communication
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No